CLINICAL TRIAL: NCT06012604
Title: Treatment of Post-radiation Xerostomia With Allogeneic Mesenchymal Stromal Stem Cells: a Pilot Study
Brief Title: Treatment of Post-radiation Xerostomia With Allogeneic Mesenchymal Stromal Stem Cells
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Oncology Ljubljana (Other)
Collaborators: Blood Transfusion Centre of Slovenia (Other Government); University Medical Centre Ljubljana (Other); University of Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERIDNPVO-0038/2023
Record Dates: First submitted 2023-08-05; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Xerostomia Following Radiotherapy
Keywords: post-radiation xerostomia; allogenic mesenchyma stromal stem cells; toxicity; effectiveness

STUDY DESIGN:
Intervention Model Description: intervention group control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- allogeneic mesenchymal stromal stem cells (Experimental): Application of allogeneic mesenchymal stromal stem cells (MSC, derived from umbilical cord tissue) under ultrasound guidance into both parotid and submandibular glands.
  Interventions: Biological: allogeneic mesenchymal stromal stem cells

INTERVENTIONS:
Biological: allogeneic mesenchymal stromal stem cells — mesenchymal stromal stem cells injection under ultrasound guidance into parotid and submandibular glands

SUMMARY:
The goal of this clinical trial is to learn about toxicity of allogeneic mesenchymal stromal stem cells (MSC, derived from umbilical cord tissue) treatment in head and neck cancer patients with for post-radiation xerostomia. The main question it aims to answer is the toxicity of intervention and the secondary objective is to assess preliminary efficacy. Participants will receive MSC in both parotid and submandibular glands: the toxicity of the intervention will be assessed using CTCAE v5.0 and its effect will be evaluated through measuring salivary flow and composition, radiologically (ultrasonography, magnetic resonance imaging), with scintigraphy and questionnaires. In the control group, salivary gland function (salivary flow and saliva composition) will be assessed for comparison with the intervention group.

DETAILED DESCRIPTION:
The aim of the study is to assess the safety and preliminary efficacy of treating xerostomia with allogeneic mesenchymal stromal stem cells (MSC) derived from umbilical cord tissue. This is a non-randomized, single-center, non-blinded Phase I study. There will be 10 patients in the intervention group and 10 healthy volunteers in the control group. In the intervention group, patients who were successfully treated with (chemo)radiotherapy for oropharyngeal squamous cell carcinoma two or more years ago and have xerostomia of grade 2 or 3 according to CTCAE v.5.0 will receive MSC injections under ultrasound guidance into both parotid and submandibular glands (1 ml syringe with 50×106 MSC and 0.5 ml syringe with 25×106 MSC). Before the application, measurements of unstimulated and stimulated saliva flow, saliva composition, and blood parameters (complete blood count, biochemical tests, prothrombin time, international normalized ratio) will be performed. Magnetic resonance imaging of the glands (to assess changes in volume, signal, and diffusivity), ultrasound elastography (to assess gland consistency), salivary gland scintigraphy with pertechnetate ([99mTc]TcO4-, to evaluate radioisotope uptake in functioning parenchyma and excretory fraction of each gland) and scintigraphy with hexamethylpropyleneamine oxime ([99mTc]Tc-HMPAO)-labeled MSC (to assess distribution, retention, and migration of MSC from the site of application) will also be conducted, along with a biopsy from one of the four glands (to evaluate morphological changes in glandular tissue). Patients will complete two xerostomia questionnaires and a quality of life questionnaire European Organization for Research and Treatment of Cancer Quality of Life H&N35. On the 1st and 5th day after the intervention (day 0), patients will be examined, and toxicity will be assessed according to CTCAE v5.0. The effect of the intervention will be evaluated at 4 weeks and 4 months, repeating the tests performed before the intervention, with the exception of the biopsy and scintigraphy, which will be repeated only 4 months after the intervention (from the same gland as the first time). In the control group, healthy individuals will submit saliva samples to determine unstimulated and stimulated saliva flow and saliva composition (for comparison with the intervention group).

ELIGIBILITY:
Inclusion Criteria:

* squamous cell carcinoma of the oropharynx, Union for International Cancer Control TNM Classification of Malignant Tumors )8th ed.) clinical stage T1-2N+ or cT3-4cN0-3 M0, treated with curative intent radiotherapy (tumor dose 66-70 Gy, bilateral neck irradiation) with or without concurrent chemotherapy
* 2 years or more post-treatment without signs of locoregional recurrence or systemic metastasis
* non-smoker or former smoker (quit smoking ≥2 years ago)
* mean radiation dose >26 Gy to each of the parotid glands and >35 Gy to each of the submandibular glands
* xerostomia of grade 2 or 3, assessed according to the CTCAE v5.0 scale
* Clinically reduced salivary flow and hyposalivation (unstimulated whole saliva flow rate 0.05-0.20 ml/min)
* age between 18-75 years
* both sexes
* signed "Informed Consent Form" for participation in the study

Exclusion Criteria:

* newly diagnosed malignancy anywhere in the body within the past two years
* active smoker
* use of medications with potential to cause dry mouth (e.g., tricyclic antidepressants, antipsychotics, decongestants, bronchodilators, antihypertensives like beta-blockers and diuretics, antihistamines, hypnotic sedatives, opioids, and muscle relaxants)
* other salivary gland diseases (e.g., Sjögren's syndrome, scleroderma, sialolithiasis, etc.)
* patients on anticoagulant therapy that cannot be discontinued during the intervention
* pregnancy or planned pregnancy within the next two years
* breastfeeding
* active, uncontrolled infection or other medical (including psychiatric) conditions that, in the researchers' opinion, do not allow for the safe administration of the planned therapy and performance of the follow-up procedures
* known substance abuse or alcoholism

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Safety: Number of patients with serious adverse events | 4 months
  Registration of number of patients with serious adverse events in a 4 months follow-up period

SECONDARY OUTCOMES:
Efficacy: Change in unstimulated and stimulated whole salivary flow rate | 4 months
  Flow rates assessed by sialometry
Efficacy: Change in saliva composition | 4 months
  Change in saliva composition
Efficacy: Change in subjective assessment of xerostomia | 4 months
  Change in subjective assessment of xerostomia evaluated by Visual Analog Scale (VAS) questionnaire
Efficacy: Change in quality of life | at baseline and 4 weeks and 4 months after intervention
  Change in quality of life evaluated by QLQ-H&N-35 questionnaire
Efficacy: performance of MSCs application | 4 months
  Assessed by salivary gland scintigraphy with [99mTc]Tc-HMPAO labeled MSCs
Efficacy: Salivary gland function | 4 months
  Assessed by salivary gland scintigraphy with pertechnetate ([99mTc]TcO4-)
Efficacy: salivary gland appearance | 4 months
  Assessed by magnetic resonance imaging and ultrasonography
Efficacy: salivary gland structure | 4 months
  Assessed by histopathological examination of salivary gland tissue sample

CONTACTS AND LOCATIONS:
Locations (4):
- Slovenia (4):
  - Blood Transfusion Center of Slovenia, Ljubljana
  - Institute of Oncology Ljubljana, Ljubljana
  - University Clinical Center Ljubljana, Ljubljana
  - University of Ljubljana, Ljubljana

IPD SHARING:
Plan to Share IPD: No